CLINICAL TRIAL: NCT00637273
Title: A Randomized, Double-Blind, Parallel-Group, Multicenter Study to Compare the Glycemic Effects, Safety, and Tolerability of Exenatide Long-Acting Release(Once Weekly) to Those of Sitagliptin and a Thiazolidinedione in Subjects With Type 2 Diabetes Mellitus Treated With Metformin
Brief Title: A Study to Compare the Glycemic Effects, Safety, and Tolerability of Exenatide Once Weekly to Those of Sitagliptin and Pioglitazone,in Subjects With Type 2 Diabetes Treated With Metformin (DURATION - 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCB106 (DURATION - 2)
Record Dates: First submitted 2008-03-06; First posted 2008-03-17 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide once weekly; Byetta; sitagliptin; Januvia; thiazolidinedione; Amylin; Lilly; Pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: exenatide once weekly; Drug: placebo tablet
- 2 (Active Comparator)
  Interventions: Drug: sitagliptin; Drug: placebo once weekly
- 3 (Active Comparator)
  Interventions: Drug: pioglitazone; Drug: placebo once weekly

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, 2.0mg, once a week
  Arms: 1
Drug: sitagliptin — oral tablet, 100mg, once a day
  Other Names: Januvia
  Arms: 2
Drug: pioglitazone — oral tablet, 45mg, once a day
  Arms: 3
Drug: placebo tablet — oral tablet, once a day
  Arms: 1
Drug: placebo once weekly — subcutaneous injection, once a week
  Arms: 2; 3

SUMMARY:
This study will compare the benefits of exenatide once weekly treatment to those achieved by the approved antidiabetic therapies sitagliptin and pioglitazone in subjects whose type 2 diabetes is managed with metformin therapy alone. The safety and tolerability of the three treatment regimens will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Has been diagnosed with type 2 diabetes mellitus
* Has a hemoglobin-specific A1c fraction (HbA1c) of 7.1% to 11.0%, inclusive, at study start
* Has a body mass index (BMI)of 25 kg/m2 to 45 kg/m2, inclusive, at study start
* Has been on a stable treatment regimen of metformin for a minimum of 2 months prior to study start
* Either is not treated with or has been on a stable treatment regimen with any of the following medications for a minimum of 2 months prior to study start:

  1. Hormone replacement therapy (female subjects)
  2. Oral contraceptives (female subjects)
  3. Antihypertensive agents
  4. Lipid-lowering agents
  5. Thyroid replacement therapy
  6. Antidepressant agents
  7. Drugs known to affect body weight, including prescription medications (e.g. orlistat [XENICAL®], sibutramine [MERIDIA®], topiramate [TOPAMAX®]) and over-the-counter antiobesity agents

Exclusion Criteria:

* Has been previously exposed to exenatide once weekly
* Has donated blood within 60 days of study start or is planning to donate blood during the study
* Currently being treated, or is expected to require or undergo treatment with any of the following treatment-excluded medications:

  1. Exenatide (BYETTA®) or any Dipeptidyl peptidase-4 DPP-4)inhibitor, sulfonylurea (SU), thiazolidinedione (TZD), or glucagon-like peptide (GLP)-1 analog within 3 months prior to study start
  2. Alpha-glucosidase inhibitor, meglitinide, nateglinide, or pramlintide (SYMLIN®) within 30 days of study start
  3. Insulin within 2 weeks of study start or for more than 1 week within 3 months of study start
  4. Systemic corticosteroids by oral, intravenous, or intramuscular route; or potent, inhaled, or intrapulmonary (including ADVAIR®) steroids known to have a high rate of systemic absorption
  5. Drugs interacting with the CYP2C8 enzyme system, including gemfibrozil (LOPID®) and rifampin
* Has received any investigational drug within 1 month (or five half-lives of investigational drug, whichever is greater) of study start
* Has previously experienced a clinically significant adverse event (e.g., significant edema) related to TZD or DPP-4 inhibitor use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (62):
- United States (51):
  - Research Site, Peoria, Arizona
  - Research Site, Artesia, California
  - Research Site, Concord, California
  - Research Site, Encino, California
  - Research Site, Greenbrae, California
  - Research Site, La Mesa, California
  - Research Site, Orange, California
  - Research Site, Walnut Creek, California
  - Research Site, Whittier, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Coral Gables, Florida
  - Research Site, DeLand, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Avon, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Paducah, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Oxon Hill, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Chelsea, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, New Hyde Park, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Durham, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Athens, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Rapid City, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
- India (5):
  - Research Site, Bangalore
  - Research Site, Indore
  - Research Site, Karnāl
  - Research Site, Mumbai
  - Research Site, Pune
- Mexico (6):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Cuernavaca, Morelos
  - Research Site, Monterrey, NuevoLeon
  - Research Site, Toluca, State of Mexico

REFERENCES:
- [Derived] Guja C, Frias JP, Suchower L, Hardy E, Marr G, Sjostrom CD, Jabbour SA. Safety and Efficacy of Exenatide Once Weekly in Participants with Type 2 Diabetes and Stage 2/3 Chronic Kidney Disease. Diabetes Ther. 2020 Jul;11(7):1467-1480. doi: 10.1007/s13300-020-00815-z. Epub 2020 Apr 18. PMID 32306296
- [Derived] Malloy J, Meloni A, Han J. Efficacy and tolerability of exenatide once weekly versus sitagliptin in patients with type 2 diabetes mellitus: a retrospective analysis of pooled clinical trial data. Postgrad Med. 2013 May;125(3):58-67. doi: 10.3810/pgm.2013.05.2661. PMID 23748507
- [Derived] Grimm M, Han J, Weaver C, Griffin P, Schulteis CT, Dong H, Malloy J. Efficacy, safety, and tolerability of exenatide once weekly in patients with type 2 diabetes mellitus: an integrated analysis of the DURATION trials. Postgrad Med. 2013 May;125(3):47-57. doi: 10.3810/pgm.2013.05.2660. PMID 23748506
- [Derived] Meloni AR, DeYoung MB, Han J, Best JH, Grimm M. Treatment of patients with type 2 diabetes with exenatide once weekly versus oral glucose-lowering medications or insulin glargine: achievement of glycemic and cardiovascular goals. Cardiovasc Diabetol. 2013 Mar 23;12:48. doi: 10.1186/1475-2840-12-48. PMID 23522121
- [Derived] Peyrot M, Bushnell DM, Best JH, Martin ML, Cameron A, Patrick DL. Development and validation of the self-management profile for type 2 diabetes (SMP-T2D). Health Qual Life Outcomes. 2012 Oct 5;10:125. doi: 10.1186/1477-7525-10-125. PMID 23039868
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Derived] Wysham C, Bergenstal R, Malloy J, Yan P, Walsh B, Malone J, Taylor K. DURATION-2: efficacy and safety of switching from maximum daily sitagliptin or pioglitazone to once-weekly exenatide. Diabet Med. 2011 Jun;28(6):705-14. doi: 10.1111/j.1464-5491.2011.03301.x. PMID 21434995
- [Derived] Bergenstal RM, Wysham C, Macconell L, Malloy J, Walsh B, Yan P, Wilhelm K, Malone J, Porter LE; DURATION-2 Study Group. Efficacy and safety of exenatide once weekly versus sitagliptin or pioglitazone as an adjunct to metformin for treatment of type 2 diabetes (DURATION-2): a randomised trial. Lancet. 2010 Aug 7;376(9739):431-9. doi: 10.1016/S0140-6736(10)60590-9. Epub 2010 Jun 26. PMID 20580422

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Once Weekly: Exenatide once weekly 2 mg subcutaneous weekly plus placebo oral once daily in the morning
- Sitagliptin: Sitagliptin 100 mg oral once daily in the morning plus placebo once weekly subcutaneous weekly
- Pioglitazone: Pioglitazone 45 mg oral once daily in the morning plus placebo once weekly subcutaneous weekly
Period: Overall Study
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Started | 170 | 172 | 172
Intent to Treat (ITT) | 160 | 166 | 165
Completed | 127 | 144 | 131
Not Completed | 43 | 28 | 41
Not completed — Adverse Event | 11 | 5 | 7
Not completed — Lost to Follow-up | 8 | 9 | 13
Not completed — Protocol Violation | 2 | 4 | 1
Not completed — Withdrawal of Consent | 18 | 6 | 18
Not completed — Investigator Decision | 1 | 3 | 1
Not completed — Administrative | 2 | 0 | 0
Not completed — Loss of Glucose Control | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone | Total
Number analyzed (Participants) | 160 | 166 | 165 | 491
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 140 | 149 | 143 | 432
  >=65 years | 20 | 17 | 22 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.41) | 52.2 (10.54) | 53.0 (9.92) | 52.5 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 80 | 86 | 237
  Male | 89 | 86 | 79 | 254
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.6 (1.20) | 8.5 (1.17) | 8.5 (1.08) | 8.5 (1.15)
Weight [Mean (Standard Deviation); unit: kg] | 89.1 (19.55) | 87.0 (20.25) | 87.9 (20.49) | 88.0 (20.08)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Absolute change in HbA1c from baseline (Day 1) to Week 26 [Week 26 - Baseline].
Time Frame: Day 1, Week 26
Population: The ITT Population included randomized subjects who received at least one injection of study medication. Missing data up to Week 26 were imputed using the last observation carried forward (LOCF) approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 159 | 162 | 160
percentage of total hemoglobin | -1.55 (0.100) | -0.92 (0.099) | -1.23 (0.099)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Null hypothesis: no difference across treatments. Alternative hypothesis: a difference exists between exenatide once weekly and at least one comparator group (sitagliptin or pioglitazone). Power: Assuming 10% dropout, delta=0.5%, and common SD=1.2%, 450 subjects would provide >90% power to detect a treatment difference (alpha=0.05, two-sided) in the change in HbA1c between exenatide once weekly and sitagliptin or pioglitazone, with Hochberg's multiplicity adjustment method; Test type: Superiority or Other; p < .0001, ANOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Analysis of Variance (ANOVA) model includes treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors; Least Squares Mean Difference = 0.63, 95% CI 2-sided [0.37 to 0.89], Standard Error of Mean 0.131
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0165, ANOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Analysis of Variance (ANOVA) model includes treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors; Least Squares Mean Difference = 0.32, 95% CI 2-sided [0.06 to 0.57], Standard Error of Mean 0.131

2. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <7% at Week 26
Description: Percentages of subjects achieving HbA1c target values of <7% at Week 26.
Time Frame: Week 26
Population: ITT Population. Missing data up to Week 26 were imputed using LOCF approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement. Subjects without post-baseline HbA1c measurement were categorized as not achieving goal.
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 160 | 166 | 165
percentage of subjects | 58.8 | 30.7 | 43.6
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Percentage of subjects achieving HbA1c target of <7% at Week 26 were compared between treatments using a Cochran Mantel Haenszel (CMH) test, in which baseline HbA1c stratum (<9% or >=9%) and country served as stratification factors. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0015, Cochran-Mantel-Haenszel — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <=6.5% at Week 26
Description: Percentages of subjects achieving HbA1c target values of <=6.5% at Week 26.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 160 | 166 | 165
percentage of subjects | 38.8 | 15.7 | 26.7
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Percentages of subjects achieving HbA1c target of <=6.5% at Week 26 were compared between treatments using a CMH test, in which baseline HbA1c stratum (<9% or >=9%) and country served as stratification factors. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0120, Cochran-Mantel-Haenszel — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons

4. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <=6.0% at Week 26
Description: Percentages of subjects achieving HbA1c target values of <=6.0% at Week 26.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 160 | 166 | 165
percentage of subjects | 13.8 | 9.0 | 4.8
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Percentages of subjects achieving HbA1c target of <=6.0% at Week 26 were compared between treatments using a CMH test, in which baseline HbA1c stratum (<9% or >=9%) and country served as stratification factors. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.1700, Cochran-Mantel-Haenszel — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0091, Cochran-Mantel-Haenszel — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons

5. Secondary Outcome: Change in Body Weight From Baseline to Week 26
Description: Change in body weight from baseline (Day 1) to Week 26.
Time Frame: Day 1, Week 26
Population: ITT Population. Missing data up to Week 26 were imputed using the LOCF approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 160 | 163 | 165
kg | -2.31 (0.323) | -0.77 (0.322) | 2.79 (0.320)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Change in body weight from baseline (Day 1) to Week 26 was analyzed by an analysis of covariance (ANCOVA) model including treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors, and baseline value of body weight as a covariate. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.0002, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 1.54, 95% CI 2-sided [0.72 to 2.35], Standard Error of Mean 0.416
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 5.10, 95% CI 2-sided [4.28 to 5.91], Standard Error of Mean 0.415

6. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 26
Description: Change in fasting plasma glucose from baseline (Day 1) to Week 26.
Time Frame: Day 1, Week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 155 | 161 | 158
mg/dL | -31.8 (3.79) | -16.3 (3.72) | -27.3 (3.75)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Change in fasting plasma glucose from baseline (Day 1) to Week 26 was analyzed using an ANCOVA model including treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors, and baseline value of fasting plasma glucose as a covariate. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.0038, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 15.5, 95% CI 2-sided [5.7 to 25.2], Standard Error of Mean 4.95
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.3729, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 4.4, 95% CI 2-sided [-5.3 to 14.2], Standard Error of Mean 4.98

7. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 26
Description: Change in systolic blood pressure from baseline (Day 1) to Week 26.
Time Frame: Day 1, Week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 160 | 163 | 165
mmHg | -3.6 (0.97) | 0.2 (0.95) | -1.6 (0.95)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Change in systolic blood pressure from baseline (Day 1) to Week 26 was analyzed by an ANCOVA model including treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors, and baseline value of systolic blood pressure as a covariate. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.0055, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 3.8, 95% CI 2-sided [1.3 to 6.3], Standard Error of Mean 1.26
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.1117, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 2.0, 95% CI 2-sided [-0.5 to 4.5], Standard Error of Mean 1.25

8. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 26
Description: Change in diastolic blood pressure from baseline (Day 1) to Week 26.
Time Frame: Day 1, Week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 160 | 163 | 165
mmHg | -1.4 (0.57) | -0.4 (0.57) | -2.5 (0.56)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Change in diastolic blood pressure from baseline (Day 1) to Week 26 was analyzed by an ANCOVA model including treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors, and baseline value of diastolic blood pressure as a covariate. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.1685, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 1.0, 95% CI 2-sided [-0.4 to 2.5], Standard Error of Mean 0.75
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.1685, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-2.6 to 0.4], Standard Error of Mean 0.75

9. Secondary Outcome: Change in Fasting Total Cholesterol From Baseline to Week 26
Description: Change in fasting total cholesterol from baseline (Day 1) to Week 26.
Time Frame: Day 1, Week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 146 | 147 | 154
mg/dL | -0.6 (2.51) | 3.1 (2.49) | 6.2 (2.46)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Change in fasting total cholesterol from baseline (Day 1) to Week 26 was analyzed by an ANCOVA model including treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors, and baseline value of fasting total cholesterol as a covariate. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.2686, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 3.7, 95% CI 2-sided [-2.8 to 10.2], Standard Error of Mean 3.31
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0814, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 6.8, 95% CI 2-sided [0.3 to 13.2], Standard Error of Mean 3.30

10. Secondary Outcome: Change in Fasting High-density Lipoprotein (HDL) From Baseline to Week 26
Description: Change in fasting HDL from baseline (Day 1) to Week 26.
Time Frame: Day 1, Week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 146 | 147 | 154
mg/dL | 2.0 (0.61) | 2.0 (0.60) | 6.2 (0.59)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Change in fasting HDL from baseline (Day 1) to Week 26 was analyzed by an ANCOVA model including treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors, and baseline value of fasting HDL as a covariate. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.9546, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = -0.0, 95% CI 2-sided [-1.6 to 1.5], Standard Error of Mean 0.80
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Least Squares Mean Difference = 4.2, 95% CI 2-sided [2.6 to 5.7], Standard Error of Mean 0.79

11. Secondary Outcome: Ratio of Fasting Triglycerides at Week 26 to Baseline
Description: Ratio of triglycerides (measured in mg/dL) at Week 26 to baseline (Day 1). Log (Postbaseline Triglycerides) - log (Baseline Triglycerides); change from baseline to endpoint is presented as ratio of endpoint to baseline.
Time Frame: Day 1, Week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 159 | 161 | 159
ratio | 0.95 (0.029) | 0.95 (0.028) | 0.84 (0.025)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Sitagliptin; Analysis: Triglycerides data were logarithm-transformed and the change at Week 26 to baseline (Day 1), expressed as the ratio, was analyzed by an ANCOVA model including treatment, country, and baseline HbA1c stratum (<9.0% or >=9.0%) as factors, and baseline value of fasting triglycerides as a covariate. Null hypothesis: no difference across treatments. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.9718, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Geometric Least Squares Mean Ratio = 1.00, 95% CI 2-sided [0.93 to 1.08], Standard Error of Mean 0.040
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.0062, ANCOVA — Adjusted p-value was derived using Hochberg's procedure for multiple treatment comparisons; Geometric Least Squares Mean Ratio = 0.89, 95% CI 2-sided [0.82 to 0.96], Standard Error of Mean 0.035

12. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Hypoglycemic Events
Description: Major hypoglycemia: events that, in the judgment of the investigator or physician, resulted in loss of consciousness, seizure, coma, or other change in mental status consistent with neuroglycopenia, in which symptoms resolved after administration of intramuscular glucagon or intravenous glucose, required third-party assistance, and was accompanied by a blood glucose concentration < 54 mg/dL prior to treatment. Minor hypoglycemia: symptoms consistent with hypoglycemia and blood glucose concentration < 54 mg/dL prior to treatment and not classified as major hypoglycemia.
Time Frame: Day 1 to Week 26
Population: ITT Population.
Measure: Mean (Standard Error); unit: rate per subject-year
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 160 | 166 | 165
rate per subject-year
  Treatment-Emergent Major Hypoglycemia | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.00)
  Treatment-Emergent Minor Hypoglycemia | 0.03 (0.021) | 0.12 (0.039) | 0.01 (0.014)

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly | Sitagliptin | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 4/160 | 5/166 | 10/165
Other Adverse Events (participants affected / at risk) | 81/160 | 59/166 | 61/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=160) | Sitagliptin (N=166) | Pioglitazone (N=165)
Cryptogenic organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Viral pericarditis (Infections and infestations) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 2
Dengue fever (Infections and infestations) | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Pancreatic abscess (Infections and infestations) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=160) | Sitagliptin (N=166) | Pioglitazone (N=165)
Nausea (Gastrointestinal disorders) | 38 | 16 | 8
Diarrhoea (Gastrointestinal disorders) | 29 | 16 | 12
Vomiting (Gastrointestinal disorders) | 18 | 4 | 5
Headache (Nervous system disorders) | 15 | 15 | 7
Urinary tract infection (Infections and infestations) | 10 | 9 | 6
Constipation (Gastrointestinal disorders) | 9 | 3 | 2
Fatigue (General disorders) | 9 | 0 | 5
Injection site pruritus (General disorders) | 8 | 8 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 15 | 17
Sinusitis (Infections and infestations) | 5 | 2 | 11
Oedema peripheral (General disorders) | 2 | 5 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less